CLINICAL TRIAL: NCT02021643
Title: A Phase 3b, Multicenter, Open-Label, Randomized Study to Investigate the Efficacy and Safety of Sofosbuvir Plus Ribavirin (± Pegylated Interferon) in Subjects With Chronic Genotype 1, 2, 3 and 6 HCV Infection
Brief Title: Efficacy and Safety of Sofosbuvir Plus Ribavirin in Adults With Chronic HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0115
Record Dates: First submitted 2013-11-26; First posted 2013-12-27 (Estimated); Results first posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2017-08

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — Sofosbuvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Sofosbuvir+RBV+PEG 12 weeks (Experimental): Participants with genotype 1 or 6 will receive sofosbuvir+RBV+Peg-IFNα-2a for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV; Drug: PEG
- Sofosbuvir+RBV 12 weeks (Experimental): Participants with genotype 1, 2 or 6 will receive sofosbuvir+RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- Sofosbuvir+RBV 16 weeks (Experimental): Participants with genotype 1, 6 will receive sofosbuvir+RBV for 16 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- Sofosbuvir+RBV 24 Weeks (Experimental): Participants with genotype 1, 3, or 6 will receive sofosbuvir+RBV for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
Drug: PEG — Pegylated interferon alfa-2a (Peg-IFNα-2a) 180 µg/0.5 mL pre-filled syringe administered subcutaneously once a week
  Other Names: Pegasys®
  Arms: Sofosbuvir+RBV+PEG 12 weeks

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety and tolerability of treatment with sofosbuvir (SOF)+ ribavirin (RBV), with or without Pegylated interferon alfa (Peg-IFNα-2a/ PEG)) in participants with chronic genotype (GT)-1, 2, 3, and 6 Hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* HCV treatment-naive (HCV genotype 1, 2, 3 or 6), defined as no prior exposure to any interferon (IFN), RBV, or other approved or experimental HCV-specific direct-acting antiviral agent, or HCV treatment-experienced (HCV genotype 1, 2, 3, or 6 only) with medical records that include sufficient detail of prior treatment with IFN to allow for categorization of prior response as either IFN Intolerant, non-responder, or experiences viral breakthrough or relapse
* HCV infection documented by anti-HCV antibody test, genotyping test, or liver biopsy

Key Exclusion Criteria:

* Current or prior history of any clinically-significant illness (other than HCV)
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non-HCV etiology
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (35):
- China (17):
  - Beijing
  - Chongqing
  - Fujian
  - Guangdong
  - Guangxi
  - Hainan
  - Hebei
  - Hubei
  - Hunan
  - Jiangxi
  - Jilin
  - Jin’an
  - Liaoyang
  - Shanghai
  - Sichuan
  - Yunnan
  - Zhejiang
- Hong Kong (2):
  - Hong Kong
  - Shatin
- South Korea (7):
  - Incheon, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Ansan-si
  - Bucheon-si
  - Busan
  - Daegu
  - Seoul
- Taiwan (7):
  - Chang-hua
  - Kaohsiung City
  - Keelung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Vietnam (2):
  - Hanoi
  - Ho Chi Minh City

REFERENCES:
- [Result] Lai CL, Wong VW, Yuen MF, Yang JC, Knox SJ, Mo H, Han LL, Brainard DM, Chan HL. Sofosbuvir plus ribavirin for the treatment of patients with chronic genotype 1 or 6 hepatitis C virus infection in Hong Kong. Aliment Pharmacol Ther. 2016 Jan;43(1):96-101. doi: 10.1111/apt.13429. Epub 2015 Oct 26. PMID 26503414
- [Result] Ahn SH, Lim YS, Lee KS, Paik SW, Lee YJ, Jeong SH, Kim JH, Yoon SK, Yim HJ, Tak WY, Han SY, Yang JC, Mo H, Mathias A, Han L, Knox SJ, Brainard DM, Kim YJ, Byun KS, Kim YS, Heo J, Han KH. A phase 3b study of sofosbuvir plus ribavirin in treatment-naive and treatment-experienced Korean patients chronically infected with genotype 2 hepatitis C virus. J Viral Hepat. 2016 May;23(5):358-65. doi: 10.1111/jvh.12499. Epub 2016 Feb 10. PMID 26864153
- [Result] Kao JH, Chien RN, Chang TT, Peng CY, Hu TH, Lo GH, Wang HY, Chen JJ, Yang JC, Knox SJ, Han L, Mo H, Mathias A, Brainard DM, Sheen IS, Hsu YC, Chu CJ, Chuang WL. A phase 3b study of sofosbuvir plus ribavirin in Taiwanese patients with chronic genotype 2 hepatitis C virus infection. Liver Int. 2016 Aug;36(8):1101-7. doi: 10.1111/liv.13082. Epub 2016 Mar 23. PMID 26835876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 61 study sites in Asia. The first participant was screened on 10 December 2013. The last study visit occurred on 03 November 2016.
Pre-assignment Details: 815 participants were screened.
Groups:
- SOF+PEG+RBV 12 Weeks: Participants with genotype 1 or 6 received Sofosbuvir (Sovaldi®; SOF) 400 mg tablet once daily + Pegylated interferon alfa-2a (PEG) 180 µg/0.5 mL pre-filled syringe administered subcutaneously once a week + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 12 Weeks: Participants with genotype 1, 2 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 16 Weeks: Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 16 weeks
- SOF+RBV 24 Weeks: Participants with genotype 1, 3 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks
Period: Overall Study
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+RBV 12 Weeks | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks
Started | 156 | 290 | 11 | 230
Completed | 147 | 280 | 11 | 218
Not Completed | 9 | 10 | 0 | 12
Not completed — Enrolled but Never Treated | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Investigator's Discretion | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 6 | 0 | 12
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least one dose of study drug.
Groups:
- SOF+PEG+RBV 12 Weeks (GT 1 and GT6): Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + PEG 180 µg/0.5 mL pre-filled syringe administered subcutaneously once a week + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 12 Weeks (GT1 and GT6): Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 16 Weeks (GT1 and GT6): Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 16 weeks
- SOF+RBV 24 Weeks (GT1 and GT6): Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks
- SOF+RBV 12 Weeks (GT2): Participants with genotype 2 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 24 Weeks (GT3): Participants with genotype 3 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks
- Total: Total of all reporting groups
Arm/Group | SOF+PEG+RBV 12 Weeks (GT 1 and GT6) | SOF+RBV 12 Weeks (GT1 and GT6) | SOF+RBV 16 Weeks (GT1 and GT6) | SOF+RBV 24 Weeks (GT1 and GT6) | SOF+RBV 12 Weeks (GT2) | SOF+RBV 24 Weeks (GT3) | Total
Number analyzed (Participants) | 155 | 10 | 11 | 104 | 280 | 126 | 686
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.8) | 43 (17.2) | 43 (17.6) | 49 (13.3) | 53 (12.3) | 40 (8.1) | 47 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 5 | 2 | 61 | 160 | 56 | 351
  Male | 88 | 5 | 9 | 43 | 120 | 70 | 335
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 155 | 10 | 11 | 104 | 280 | 126 | 686
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 151 | 10 | 11 | 98 | 280 | 126 | 676
  Not Disclosed | 4 | 0 | 0 | 6 | 0 | 0 | 10
Region of Enrollment [Number; unit: participants]
  China | 130 | 0 | 0 | 69 | 64 | 126 | 389
  Hong Kong | 0 | 10 | 11 | 10 | 0 | 0 | 31
  South Korea | 0 | 0 | 0 | 0 | 129 | 0 | 129
  Taiwan | 0 | 0 | 0 | 0 | 87 | 0 | 87
  Vietnam | 25 | 0 | 0 | 25 | 0 | 0 | 50
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 108 | 7 | 7 | 81 | 0 | 0 | 203
  Genotype 2 | 0 | 0 | 0 | 0 | 280 | 0 | 280
  Genotype 3 | 0 | 0 | 0 | 0 | 0 | 126 | 126
  Genotype 6 | 47 | 3 | 4 | 23 | 0 | 0 | 77
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 114 | 8 | 11 | 74 | 237 | 102 | 546
    CT | 40 | 2 | 0 | 29 | 42 | 23 | 136
    TT | 1 | 0 | 0 | 1 | 1 | 1 | 4
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.74) | 6.3 (0.49) | 6.2 (0.88) | 6.5 (0.71) | 6.2 (0.96) | 6.2 (0.71) | 6.3 (0.84)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 21 | 2 | 6 | 22 | 87 | 32 | 170
  ≥ 800,000 IU/mL | 134 | 8 | 5 | 82 | 193 | 94 | 516

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 is defined as HCV RNA < the lower limit of quantification (LLOQ; ie, < 25 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who enrolled in the study and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks (GT 1 and GT6) | SOF+RBV 12 Weeks (GT1 and GT6) | SOF+RBV 16 Weeks (GT1 and GT6) | SOF+RBV 24 Weeks (GT1 and GT6) | SOF+RBV 12 Weeks (GT2) | SOF+RBV 24 Weeks (GT3)
Number analyzed (Participants) | 155 | 10 | 11 | 104 | 280 | 126
percentage of participants | 95.5 [90.9 to 98.2] | 100 [69.2 to 100] | 100 [71.5 to 100] | 94.2 [87.9 to 97.9] | 96.8 [94.0 to 98.5] | 95.2 [89.9 to 98.2]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- SOF+PEG+RBV 12 Weeks: Participants with genotype (GT) 1 or 6 received SOF 400 mg tablet once daily + PEG 180 µg/0.5 mL pre-filled syringe administered subcutaneously once a week + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 16 Weeks: Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+RBV 12 Weeks | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 155 | 290 | 11 | 230
Participants | 1 | 1 | 0 | 2

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 are defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+PEG+RBV 12 Weeks (GT 1 and GT6) | SOF+RBV 12 Weeks (GT1 and GT6) | SOF+RBV 16 Weeks (GT1 and GT6) | SOF+RBV 24 Weeks (GT1 and GT6) | SOF+RBV 12 Weeks (GT2) | SOF+RBV 24 Weeks (GT3)
Number analyzed (Participants) | 155 | 10 | 11 | 104 | 280 | 126
percentage of participants
  SVR4 | 96.8 [92.6 to 98.9] | 100 [69.2 to 100.0] | 100 [71.5 to 100.0] | 94.2 [87.9 to 97.9] | 97.5 [94.9 to 99.0] | 97.6 [93.2 to 99.5]
  SVR24 | 95.5 [90.9 to 98.2] | 100 [69.2 to 100.0] | 90.9 [58.7 to 99.8] | 94.2 [87.9 to 97.9] | 96.8 [94.0 to 98.5] | 95.2 [89.9 to 98.2]

4. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Failure
Description: Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment.
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+PEG+RBV 12 Weeks (GT 1 and GT6) | SOF+RBV 12 Weeks (GT1 and GT6) | SOF+RBV 16 Weeks (GT1 and GT6) | SOF+RBV 24 Weeks (GT1 and GT6) | SOF+RBV 12 Weeks (GT2) | SOF+RBV 24 Weeks (GT3)
Number analyzed (Participants) | 155 | 10 | 11 | 104 | 280 | 126
Participants | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+PEG+RBV 12 Weeks (GT 1 and GT6) | SOF+RBV 12 Weeks (GT1 and GT6) | SOF+RBV 16 Weeks (GT1 and GT6) | SOF+RBV 24 Weeks (GT1 and GT6) | SOF+RBV 12 Weeks (GT2) | SOF+RBV 24 Weeks (GT3)
Number analyzed (Participants) | 155 | 10 | 11 | 104 | 280 | 126
Participants | 7 | 0 | 0 | 6 | 6 | 6

6. Secondary Outcome: Change From Baseline in HCV RNA (log10 IU/mL)
Time Frame: Up to 24 weeks
Population: Participants in the Full Analysis Set with available data were analyzed
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+PEG+RBV 12 Weeks (GT 1 and GT6) | SOF+RBV 12 Weeks (GT1 and GT6) | SOF+RBV 16 Weeks (GT1 and GT6) | SOF+RBV 24 Weeks (GT1 and GT6) | SOF+RBV 12 Weeks (GT2) | SOF+RBV 24 Weeks (GT3)
Number analyzed (Participants) | 155 | 10 | 11 | 104 | 280 | 126
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 155 | 10 | 11 | 104 | 278 | 125
  Change at Week 1 | -4.81 (0.653) | -4.59 (0.359) | -4.36 (0.560) | -4.61 (0.607) | -4.46 (0.815) | -4.52 (0.695)
  Change at Week 2: number analyzed (Participants) | 154 | 10 | 11 | 103 | 280 | 126
  Change at Week 2 | -5.11 (0.734) | -4.89 (0.488) | -4.79 (0.858) | -5.04 (0.682) | -4.78 (1.008) | -4.86 (0.706)
  Change at Week 4 | -5.12 (0.738) | -4.89 (0.488) | -4.82 (0.880) | -5.12 (0.710) | -4.81 (1.025) | -4.87 (0.713)
  Change at Week 6 | -5.12 (0.738) | -4.89 (0.488) | -4.82 (0.880) | -5.12 (0.710) | -4.80 (1.038) | -4.87 (0.713)
  Change at Week 8: number analyzed (Participants) | 155 | 10 | 11 | 103 | 279 | 126
  Change at Week 8 | -5.12 (0.738) | -4.89 (0.488) | -4.82 (0.880) | -5.12 (0.708) | -4.83 (0.966) | -4.87 (0.713)
  Change at Week 10: number analyzed (Participants) | 155 | 10 | 11 | 103 | 279 | 126
  Change at Week 10 | -5.12 (0.738) | -4.89 (0.488) | -4.82 (0.880) | -5.12 (0.708) | -4.83 (0.966) | -4.87 (0.713)
  Change at Week 12: number analyzed (Participants) | 154 | 10 | 11 | 103 | 278 | 126
  Change at Week 12 | -5.12 (0.739) | -4.89 (0.488) | -4.82 (0.880) | -5.12 (0.708) | -4.83 (0.966) | -4.84 (0.779)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 11 | 103 | 0 | 126
  Change at Week 16 |  |  | -4.82 (0.880) | -5.12 (0.708) |  | -4.87 (0.713)
  Change at Week 20: number analyzed (Participants) | 0 | 0 | 0 | 102 | 0 | 126
  Change at Week 20 |  |  |  | -5.14 (0.701) |  | -4.87 (0.713)
  Change at Week 24: number analyzed (Participants) | 0 | 0 | 0 | 102 | 0 | 126
  Change at Week 24 |  |  |  | -5.14 (0.701) |  | -4.87 (0.713)

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks Plus 30 Days
Groups:
- SOF+PEG+RBV 12 Weeks: Participants with genotype 1 or 6 received SOF 400 mg tablet once daily + PEG 180 µg/0.5 mL pre-filled syringe administered subcutaneously once a week + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Arm/Group | SOF+PEG+RBV 12 Weeks | SOF+RBV 12 Weeks | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 5/155 | 7/290 | 0/11 | 4/230
Other Adverse Events (participants affected / at risk) | 145/155 | 215/290 | 5/11 | 177/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+PEG+RBV 12 Weeks (N=155) | SOF+RBV 12 Weeks (N=290) | SOF+RBV 16 Weeks (N=11) | SOF+RBV 24 Weeks (N=230)
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+PEG+RBV 12 Weeks (N=155) | SOF+RBV 12 Weeks (N=290) | SOF+RBV 16 Weeks (N=11) | SOF+RBV 24 Weeks (N=230)
Anaemia (Blood and lymphatic system disorders) | 30 | 22 | 1 | 27
Leukopenia (Blood and lymphatic system disorders) | 30 | 2 | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 27 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 8 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 14 | 0 | 2
Vomiting (Gastrointestinal disorders) | 6 | 8 | 1 | 1
Asthenia (General disorders) | 21 | 8 | 0 | 9
Fatigue (General disorders) | 24 | 21 | 0 | 20
Malaise (General disorders) | 0 | 3 | 2 | 1
Non-cardiac chest pain (General disorders) | 8 | 0 | 0 | 4
Pain (General disorders) | 9 | 0 | 0 | 5
Pyrexia (General disorders) | 56 | 4 | 0 | 10
Nasopharyngitis (Infections and infestations) | 6 | 21 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 11 | 30 | 2 | 27
Alanine aminotransferase increased (Investigations) | 10 | 0 | 0 | 6
Blood bilirubin increased (Investigations) | 7 | 7 | 0 | 34
Haemoglobin decreased (Investigations) | 23 | 9 | 0 | 20
Neutrophil count decreased (Investigations) | 38 | 1 | 0 | 1
Platelet count decreased (Investigations) | 37 | 1 | 0 | 2
Red blood cell count decreased (Investigations) | 11 | 6 | 0 | 16
Reticulocyte count increased (Investigations) | 13 | 15 | 0 | 35
White blood cell count decreased (Investigations) | 33 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 4 | 0 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 14 | 0 | 1
Dizziness (Nervous system disorders) | 14 | 17 | 0 | 11
Headache (Nervous system disorders) | 24 | 34 | 0 | 14
Insomnia (Psychiatric disorders) | 6 | 29 | 0 | 26
Irritability (Psychiatric disorders) | 1 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 18 | 0 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 0 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 33 | 0 | 8
Rash (Skin and subcutaneous tissue disorders) | 11 | 18 | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years